CLINICAL TRIAL: NCT06180460
Title: Managing Distress in Malignant Brain Cancer - Phase IIc RCT
Brief Title: CALM: Managing Distress in Malignant Brain Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23-20816
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Brain Tumor; Brain Metastases; Brain Cancer; Metastatic Lung Cancer; Metastatic Breast Cancer; Metastatic Melanoma; Metastatic Colon Cancer; Metastatic Kidney Cancer
Keywords: Service Members; Veterans
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Breast Neoplasms; Melanoma; Colonic Neoplasms; Kidney Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Cancer and Living Meaningfully (CALM) (Experimental): CALM optimally consists of six individual sessions of 45 to 60 minutes, delivered over a three- to six-month period. CALM sessions address four broad and interrelated domains found to be important and relevant in this population: (1) symptom management and communication with healthcare providers, (2) changes in personal relationships, (3) sense of meaning and purpose, and (4) the future, hope and mortality.
  Interventions: Behavioral: CALM
- Treatment as Usual (TAU) (Placebo Comparator): Treatment as usual (TAU) for managing distress in brain cancer involves being provided a list of local / national resources (e.g., psychologist, social worker, or other mental health providers) if an individual chooses to seek treatment for the distress they are experiencing.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: CALM — The CALM intervention is a supportive-expressive therapy that is administered by CALM trained clinicians in a particular style.
  Arms: Managing Cancer and Living Meaningfully (CALM)
Behavioral: Treatment as usual — Treatment as usual includes a list of local / national resources (e.g., psychologist, social worker, or other mental health providers) if an individual chooses to seek treatment for the distress they are experiencing.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The purpose of this study is to test an empirically supported psychotherapeutic intervention, Managing Cancer and Living Meaningfully (CALM), compared to treatment as usual (TAU) in those with malignant brain cancer diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of brain metastasis (bMET) or a malignant primary brain tumor (PBT; specifically grade III or IV and CNS diffuse large B cell lymphomas)*
* At least 2-weeks post-surgical resection or biopsy of the brain (if applicable)
* Score > 20 on the TICS
* Reported elevated depression (PHQ-9 score ≥ 10) OR death anxiety symptoms (DADDS score ≥ 15)
* Ability to read, speak, and understand English
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Major communication difficulties which would prohibit the psychotherapeutic interaction
* Inability to meet with the interventionist via an electronic device for telehealth intervention sessions
* Inability to understand and provide informed consent
* Prisoners
* Medical, psychological, or social condition that, in the opinion of the principal investigator, may increase the participant's risk of adverse events and/or prohibit the individual's participation in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of the CALM intervention- Screening Rate | Day 0
  Percent of interested individuals who undergo screening
Assess the feasibility of the CALM intervention- Consent Rate | Day 0
  Percent of eligible individuals who consent to the trial
Assess the feasibility of the CALM intervention- Intervention Retention Rate | 3 months
  Percent of consented individuals who complete the CALM intervention
Assess the feasibility of the CALM intervention- Post-Intervention Questionnaire Completion Rate | 3 months
  Percent of consented individuals who complete post-intervention questionnaires
Assess the feasibility of the CALM intervention- Follow-up Questionnaire Completion Rate | 6 months
  Percent of consented individuals who complete follow-up questionnaires
Assess the acceptability of the CALM intervention- Participant Satisfaction | 4 months
  Satisfaction ratings from participants during exit interview (e.g., Rate your overall benefit on a scale of 1-5).
Assess the acceptability of the CALM intervention- Participant Recommendation Ratings | 4 months
  Percent of participants who would recommendation CALM to others will be assessed during the exit interview (e.g., Would you recommend this program to others?)

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States